CLINICAL TRIAL: NCT06749561
Title: A Comparative Investigation of Efficacy and Complications in Light and Deep Chemical Peels
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHS/Batch-Spring23/057
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Peeling Skin Syndrome
MeSH Terms: conditions — Peeling Skin Syndrome | interventions — Chromosomes, Human, 1-3

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Group 1 — To Compare the safety and effectiveness of boyh types

SUMMARY:
Chemical peeling involves applying substances to the skin to induce controlled damage, which promotes the regeneration of fresh skin cells and enhances the skin's appearance.

DETAILED DESCRIPTION:
This study will be a cross-sectional analysis with a sample size of 112 patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females aged 18-35 years.
* Willing to provide informed consent and follow the treatment protocol.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Active skin conditions (e.g., acne, eczema).
* Use of medications that affect skin healing.
* Known allergies to chemical peel substances.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: To check the outcomes of Efficacy and Complications in Light and Deep Chemical Peels
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Dermatological Assessment Score (DAS) | 12 Months
  The area-wise percentage involvement of the involved sites is calculated as: 1 = less than 10% area; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; and 6 = more than 90%. The maximum score of PASI is 72. PASI 75 is a 75% reduction of baseline PASI score.

CONTACTS AND LOCATIONS:
Locations (1):
- Block E3 E-3 Gulberg III, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No